CLINICAL TRIAL: NCT06995859
Title: Amalgam Restorations Teaching in Pediatric Dentistry in Egyptian Universities: A Cross-sectional Study
Brief Title: Amalgam Restorations Teaching in Pediatric Dentistry
Status: Enrolling by invitation | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmin Mohamed Yousry, associate professor of pediatric dentistry, Cairo University
Other Study IDs: dental education of amalgam
Record Dates: First submitted 2025-05-08; First posted 2025-05-30 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Dental Amalgam
Keywords: dental education; amalgam restoration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric dentistry educators in Egyptian universities

SUMMARY:
To assess the pediatric dentistry educator's perception about teaching and using dental amalgam as restoration for primary teeth.

DETAILED DESCRIPTION:
Dental education has long emphasized the development of clinical skills necessary for restorative procedures. Among these, amalgam restorations have been a foundational component of dental curricula for decades due to their durability, cost-effectiveness, and historical prominence in restorative dentistry. However, in recent years, the use of amalgam has become a subject of debate due to environmental concerns related to mercury content, alongside the increasing popularity of composite materials.

To our knowledge no current data is available regarding teaching amalgam in pediatric dentistry in Egyptian dental universities. So, the aim of this study is to assess the pediatric dentistry educator's perception about teaching and using dental amalgam as restoration for primary teeth. This could help in making improvements to the dental education system ensuring that future dentists are equipped to offer patients the best treatment options based on individual needs, improving overall oral health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants included will be Pediatric dentistry educators in Egyptian universities with at least one year experience.

Exclusion Criteria:

* Pediatric dentistry educators who are not willing to participate or to complete the questionnaire will be excluded also administrative and non-teaching staff

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pediatric dentistry educators in Egyptian universities with at least one year experience.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Pediatric dentistry educator's perception about teaching amalgam restorations | 1 month
  The proportion of pediatric dentistry educator's who agree or disagree that amalgam restorations should remain part of clinical teaching for both undergraduate and postgraduate students in dental universities the outcome will be measured by questionnaire

SECONDARY OUTCOMES:
Pediatric dentistry educator's experience and confidence about using dental amalgam as restoration for primary teeth | 1 month
  The proportion of pediatric dentistry educator's who agree or disagree about using dental amalgam as restoration for primary teeth the outcome will be measured using questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol